CLINICAL TRIAL: NCT05782647
Title: Feasibility of Blood Pressure Measurement With a Wearable (Watch-type) Monitor in Patients With Syncope
Brief Title: Wearable Monitor in Patients With Syncope
Acronym: Watch-VD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09C128
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Syncope, Vasovagal
Keywords: Syncope; tilt testing; blood pressure monitoring
MeSH Terms: conditions — Syncope, Vasovagal; Syncope

STUDY DESIGN:
Intervention Model Description: Cuffless (watch type) BP monitor and standard beat-to-beat monitoring device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuffless BP monitoring (Experimental): Investigational device Omron HeartGuide® 6410T
  Interventions: Device: HeartGuide cuffless BP monitor
- Beat-to-beat BP monitoring (Active Comparator): Continuous finger BP monitoring (Finometer®, Finapres Medical Systems, Enchede, The Netherlands, and Task Force® monitor, CNSystem, Graz, Austria), based on the photoplethysmographic volume clamp method
  Interventions: Device: HeartGuide cuffless BP monitor

INTERVENTIONS:
Device: HeartGuide cuffless BP monitor — Wearable (watch-type) monitor: HeartGuide 6410T (Omron Healthcare, Kyoto, Japan)

SUMMARY:
The main purpose of this study is to assess the reliability of a new patient's self-administered wearable watch-type BP monitor in detecting episodes of hypotensive (pre)syncope. Secondary aim regards the estimation of feasibility of this tool.

DETAILED DESCRIPTION:
Background While ECG monitoring is a reliable and established method that allows to document bradycardia in a substantial proportion of patients affected by cardioinhibitory reflex syncope, the documentation of a transient hypotension is only seldom achieved in patients affected by hypotensive syncope. Conventional ambulatory blood pressure (BP) monitoring (ABPM) has important limitations due to the short period of monitoring (usually 24-48 hours) and the intermittent nature of BP measurements (usually every 15-20 min).

The main purpose of this study is to assess the reliability of a new patient's self-administered wearable watch-type BP monitor in detecting episodes of hypotensive (pre)syncope. Secondary aim regards the estimation of feasibility of this tool.

Method The study is a prospective intrapatient comparison during tilt testing between BP measured by mean of a wearable watch-type BP monitor (Omron HeartGuide 6410T, Omron Healthcare, Kyoto, Japan) and by mean of the standard methods for continuous finger BP monitoring (Finometer®, Finapres Medical Systems, Enchede, The Netherlands, and Task Force® monitor, CNSystem, Graz, Austria), based on the photoplethysmographic volume clamp method .

Study design BP values observed during tilt testing baseline and at the time of impeding syncope will be measured by mean of the HeartGuide device and will be compared with the standard of reference of BP. BP will be recorded at rest at baseline, shortly after upright in tilting position (at stabilization), at the time of occurrence of impeding syncope (presyncope) or, alternatively at the time of maximum hypotensive effect, if syncope will not occur, and finally in the recovery period at the end of the test after returning in supine position.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients,
* >18 years of age, referred for tilt testing because affected by suspected reflex syncope

Exclusion Criteria:

* Arrhythmias or the inability of HeartGuide to measure BP supine at rest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
BP during event during tilt testing | 2 hours
  Difference between baseline (rest) BP and BP at the presyncopal event ("Delta BP slope") during tilt testing with HeartGuide and with control

SECONDARY OUTCOMES:
Compliance | 2 hours
  Number of patients who will show failure of HeartGuide to measure BP during tilt event

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request to the principal investigator
Supporting Information: CSR
Time Frame: Aafter publication of the princiapl study
Access Criteria: m.brignole@auxologico.it